CLINICAL TRIAL: NCT04099654
Title: The Effect of Structured Core Stabilization Exercise Program on Functional Capacity, Physical Fitness and Quality of Life in Obese Subjects Awaiting Bariatric Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Core Stabilization Exercise Program in Obese Subjects Awaiting Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Assist.Prof.Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04/07/2019-101631
Record Dates: First submitted 2019-07-24; First posted 2019-09-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obese; Exercise; Bariatric Surgery Candidate
Keywords: obese; core stabilization; bariatric surgery; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core-Stabilization Exercise (Experimental)
  Interventions: Other: Core-Stabilization Exercise
- Counseling of physical activity (Experimental)
  Interventions: Other: Counseling of physical activity

INTERVENTIONS:
Other: Core-Stabilization Exercise — A program consisting of core stabilization exercises and physical activity counseling accompanied by physiotherapists will be applied to the study group.
  Arms: Core-Stabilization Exercise
Other: Counseling of physical activity — Only physical activity counseling will be given to the subjects in this group.
  Arms: Counseling of physical activity

SUMMARY:
In this study, our primary aim is to investigate the effects of structured core stabilization exercise program on functional capacity, body composition, muscle strength, endurance, balance, quality of life in adult obese individuals expecting bariatric surgery. Our secondary aim is to provide the individual with exercise habits and increase the level of physical activity in daily life with the exercise program planned according to the needs of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-65
* BMI ≥30 kg/m2, individuals waiting bariatric surgery
* No surgical operation in the last 6 months

Exclusion Criteria:

* Musculoskeletal disorders or systemic diseases that may prevent exercise
* The presence of psychiatric or neurological disease affecting cooperation and cognitive functions
* Presence of acute pain
* Heart pain
* Presence of previous myocardial infarction, subjective heart failure, uncontrolled diabetes and hypertension
* Regular exercise for 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Change from baseline to 8 weeks, follow up at two months
  The Six Minute Walk Test was conducted according to a standardized protocol, using an internal hallway with the 30-meter distance marked by colored tape on the floor. Participants will be told that "the purpose of this test is to see how far you can walk in six minutes." Then, they will be instructed to "walk from end to end of the hallway at your own pace, in order to cover as much ground as possible." Participants will be allowed to stop and rest during the test, but will be instructed to resume walking as soon as they were able to do so. Before the walk started and at the end of the 6-min walk, participants will be shown a modified Borg dyspnea scale printed on a card and asked to "indicate your current degree of shortness of breath" on a scale of "0 = nothing at all" to "10 = very, very severe." At the end of the walk, they will be asked if they had experienced any of the following specific symptoms: dyspnea, chest pain, light-headedness, or leg pain, or any other symptoms.
Assessment of Core Stabilization | Change from baseline to 8 weeks, follow up at two months
  Core stabilization evaluation will be done with Anterior and Side Abdominal Strength Tests, Trunk Flexor Test and Modified Push Up Test. These tests will be performed using a 2 kilogram medicine ball. Test positions are supine and sitting position.

SECONDARY OUTCOMES:
Bioelectrical Impedance Analysis-obesity score | Change from baseline to 8 weeks, follow up at two months
  Body components such as body fat percentage, body fat amount, lean body percentage, lean body mass, body water percentage, body water quantity, body mass index are calculated with bioelectrical impedance analysis. The muscle, fat and water ratio of the cases will be evaluated with Tanita Bioelectric Impedance Device. When the device assess the body fat percentage, body fat amount, lean body percentage, lean body mass, body water percentage, body water quantity and body mass index, it offers to us a score as called obesity score.
Biodex Balance System-Fall Risk Test | Change from baseline to 8 weeks, follow up at two months
  Biodex Balance System is a system that offers the possibility of evaluating the balance statically and dynamically. It is a system that measures the displacements in the center of gravity of a patient standing on an outpatient balance platform and the reactions of the support surface when the surface changes. For the static balance will be assessed with "Fall Risk Test " by using Biodex Balance system. Fall risk test offers to us a total score.
Obesity Specific Quality of Life Scale | Change from baseline to 8 weeks, follow up at two months
  Quality of life (QoL) will be measured using the Obesity Specific Quality Of Life (OSQOL) questionnaire. This disease-specific questionnaire includes 11 questions grouped into four dimensions: 1- "Physical state" (7 questions), 2- "Vitality, desire to do things" (2 questions), 3- "Relations with other people" (1 question), 4- "Psychological state" (1 question). Each question offered five possible answers ('absolutely false', 'fairly false', 'neither true nor false', 'fairly true' and 'absolutely true'), classified according to reduced QoL. For dimensions 1 and 2, a quantitative score is calculated (0% minimal QoL, 100% maximal QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No